CLINICAL TRIAL: NCT06243094
Title: Survey on Antibiotic Therapy Practices for Ventilator-Associated Pneumonia in ICU Patients
Brief Title: Antibiotic Therapy Practices for Ventilator-Associated Pneumonia (PETUNIA)
Acronym: PETUNIA
Status: Recruiting | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A01492-43
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Ventilator Associated Pneumonia
Keywords: antibiotic; intensive care; guidelines; outcome
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- microbiologically confirmed VAP: patients who meet ATS/IDSA 2005 VAP criteria with microbiological confirmation
  Interventions: Drug: Antibiotic
- non microbiologically confirmed VAP: patients who do not meet ATS/IDSA 2005 criteria with microbiological confirmation
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — All antibiotic therapy characteristics are monitored.
  Other Names: antimicrobial therapy

SUMMARY:
The French Society of Intensive Care conducts a comprehensive assessment of current antibiotic therapy practices in critically ill patients suspected of Ventilator-Associated Pneumonia (VAP).

DETAILED DESCRIPTION:
This prospective observational multicenter study will be conducted in intensive care units (ICU) across France and French-speaking regions. The primary objective of this study is to delineate the characteristics of antibiotic treatments administered for a first episode of suspected VAP. Secondary objectives include describing the outcomes of enrolled patients, assessing adherence to European guidelines regarding empirical antibiotic treatment, and identifying factors associated with mortality in patients with microbiologically confirmed VAP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the ICU
* Intubation and duration of invasive mechanical ventilation > 48 hours
* Initiation of new antibiotic therapy to treat a first suspicion of Ventilator-Associated Pneumonia (VAP)

Exclusion Criteria:

* Presence of a decision to limit active therapeutic measures at the time of initiating antibiotic therapy
* Organ donor
* Prior inclusion in the study during a previous stay in the intensive care unit (a patient cannot be included multiple times)
* Participation in an interventional study focusing on the management of VAP and directly impacting antibiotic therapy practices
* Patient and/or family opposition to participation
* Lack of affiliation with a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be ICU patients, undergoing invasive mechanical ventilation > 48h, for whom antibiotic therapy is initiated to treat a suspicion of Ventilator-Associated Pneumonia (VAP).
Sampling Method: Non-Probability Sample
Enrollment: 1060 (Estimated)
Dates: Start 2024-03-12 (Estimated); Primary Completion 2025-03-12 (Estimated); Study Completion 2025-03-12 (Estimated)

PRIMARY OUTCOMES:
Characteristics of Initial Antibiotic Treatment | 3 days
  Empirical / guided / directly targeted Monotherapy or combination therapy Monotherapy or combination therapy against resistant GNB Addition of an antibiotic active against Methicillin-Resistant Staphylococcus aureus Molecule(s) and class(es) of antibiotics Time from the onset of suspected VAP to initiation of initial antibiotic treatment Total dose in the first 24 hours for each molecule Administration modalities in the first 24 hours for each molecule Conducting plasma level measurements Appropriate treatment (in patients with microbiologically confirmed VAP) Time from the onset of suspected VAP to initiation of appropriate antibiotic treatment (in patients with microbiologically confirmed VAP)
  Note for the reviewer: our study is descriptive, and multiple characteristics of initial antibiotic treatment have been validated by the institutional review board and methodologist, as a descriptive outcome.
Characteristics of Definitive Antibiotic Treatment (for patients alive at Day 3 only) | 7 days
  Monotherapy or combination therapy Molecule(s) and class(es) of antibiotics Broadening of antibiotic spectrum Discontinuation of all antibiotics (prescribed for VAP treatment) at Day 3 and Day 5 Antibiotic de-escalation at Day 3 and Day 5 by reducing the spectrum of an initial antibiotic or by discontinuing a component of an initial combination of antibiotics
  Note for the reviewer: our study is descriptive, and multiple characteristics of definite antibiotic treatment have been validated by the institutional review board and methodologist, as a descriptive outcome.
Total Duration of Appropriate Treatment | ICU stay (up to 28 days)
  Total Duration of Appropriate Treatment for the episode of VAP

CONTACTS AND LOCATIONS:
Overall Officials: Anahita Rouzé, MD, Principal Investigator — French Intensive Care Society
Locations (1):
- Lille university hospital, Lille, Haut de France, France

IPD SHARING:
Plan to Share IPD: Undecided